CLINICAL TRIAL: NCT04535297
Title: Consequences of the COVID-19 Lockdown on Health and Well-being of Patients With Parkinson Disease and Post-stroke
Status: Completed | Type: Observational
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Galit Yogev-Seligmann, Dr., University of Haifa
Other Study IDs: 203/20
Record Dates: First submitted 2020-08-31; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Parkinson Disease; Stroke
MeSH Terms: conditions — Parkinson Disease; Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: exposure — Exposure to social distancing due to COVID-19

SUMMARY:
The study aimed at describing the effects of the COVID-19 social distancing on function, health and well-being of patients with Parkinson's disease or post-stroke, and test the association between the patient activation level and these effects.An anonymous survey was distributed through social media and patient associations.Community-living patients with Parkinson's disease or post-stroke were invited to answer the survey.

DETAILED DESCRIPTION:
People with chronic diseases like Parkinson's disease or post-stroke rely on routine medical and rehabilitative care to maintain daily function and health. These are important aspects of self-management. However, this was challenged by the social distancing due to COVID-19, which limited participation in regular routines.

The study objectives were: To (1) describe the effects of the COVID-19 social distancing on function, health and well-being of patients with Parkinson's disease or post-stroke, and (2) test the association between the patient activation level and these effects.

Community-living patients with Parkinson's disease or post-stroke were invited to answer an anonymous survey through social media and patient associations. Part 1 included 27 multiple-choice questions regarding current status and changes in function, health, medical care and well-being. Part 2 consisted of the Patient Activation Measure, describing people's knowledge, skill, and confidence in managing their own health.

ELIGIBILITY:
Inclusion Criteria:

* People diagnosed with Parkinson's disease or their caregivers, or people post-stroke or their caregivers
* Live in the community
* If a family member or caregiver completed the survey, we asked them to answer in reference to the patient.

Exclusion Criteria:

* diagnosis of COVID-19
* hospitalization in the last 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with PD or their caregivers, or patients post-stroke or their caregivers
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2020-05-10 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM®) | 1 hour
  The PAM is a self-reported validated, licensed tool to measure a patient's knowledge, skills and confidence for self-management. The overall score captures the extent to which people feel engaged and confident in taking care of their health condition. It consists of 13 statements rated on a Likert scale according to agreement. Scores are divided into 4 levels, where 1 represents patients who tend to be passive and feel overwhelmed managing their own health, and 4 represents patients who have effectively adopted self-management behaviors. We used a validated licensed Hebrew and version of the PAM supplied by Insignia Health (https://www.insigniahealth.com/products/pam-survey), which holds the copyright to the questionnaire.
Answers to multiple-choice questions | 1 hour
  participants were asked to answer 27 multiple-choice questions regarding status and change in status of mobility, mood (depression, anxiety), tiredness, social support, body weight, physical activity, rehabilitative treatments and disease symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Galit Yogev-Seligmann, Principal Investigator — University of Haifa
Locations (1):
- Galit Yogev-Seligmann, Haifa, Please Select..., Israel

IPD SHARING:
Plan to Share IPD: No